CLINICAL TRIAL: NCT02223013
Title: Relative Bioavailability and Tolerability of Two New Different Extended Release Capsules of 50 mg BIBV 308 SE Each, Versus a Solution of 50 mg BIBV 308 SE Administered Orally Twice a Day for 3.5 Days to Healthy Subjects (Cross-over, Open, Randomized)
Brief Title: Relative Bioavailability and Tolerability of Two New Different Extended Release Capsules of BIBV 308 SE, Versus a Solution of BIBV 308 SE in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 528.204
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (3):
- BIBV 308 SE solution (Active Comparator)
  Interventions: Drug: BIBV 308 SE solution
- BIBV 308 SE capsule L (Experimental)
  Interventions: Drug: BIBV 308 SE capsule L
- BIBV 308 SE capsule S (Experimental)
  Interventions: Drug: BIBV 308 SE capsule S

INTERVENTIONS:
Drug: BIBV 308 SE solution
  Arms: BIBV 308 SE solution
Drug: BIBV 308 SE capsule L
  Arms: BIBV 308 SE capsule L
Drug: BIBV 308 SE capsule S
  Arms: BIBV 308 SE capsule S

SUMMARY:
Comparative pharmacokinetics and tolerability of two experimental extended release formulations and a standard formulation of BIBV 308 SE following multiple doses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that were previously entered in at least one BIBV 308 SE study to ensure that it is known how these subjects absorb BIBV 308 SE
* Healthy subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age >= 18 and <= 55 years
* Broca >= -20% and <= +20 %

Exclusion Criteria:

* Poor individual absorption kinetics of BIBV 308 SE in previous studies
* Any findings of the medical examination (including blood pressure, pulse rate and Electrocardiogram (ECG)) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal (including thyroid) disorders
* Surgery of the gastro-intestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or acute relevant infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Hypersensitivity to BIBV 308 SE and any of the excipients
* Intake of drugs with a long half-life (> 24 hours) <= 1 month prior to administration or during the trial
* Use of any drugs which might influence the results of the trial <= 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug <= 2 months days prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking during the period of the study
* Known alcohol (> 60 g/day) or drug abuse
* Blood donation (<= 1 month prior to administration)
* Excessive physical activities (<= 5 days prior to administration)
* Any laboratory value outside the normal range of clinical relevance
* History of haemorrhagic diathesis
* History of gastro-intestinal ulcer, perforation or bleeding
* History of bronchial asthma

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 1999-04; Primary Completion 1999-05 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma at steady state (AUCss) | up to 84 hours
Maximum plasma concentration at steady state (Cmax,ss) | up to 84 hours
Minimum plasma concentration at steady state (Cmin,ss) | up to 84 hours

SECONDARY OUTCOMES:
Percent peak-to-trough fluctuation (%PTF) | up to 84 hours
Time to maximum plasma concentration in steady state (tmax,ss) | up to 84 hours
Mean residence time in steady state (MRT,ss) | up to 84 hours
Total plasma clearance (CL/f) | up to 84 hours
Quotient of Cmax,ss and AUCss (Cmax,ss/AUCss) | up to 84 hours
Number of patients with adverse events | up to 5 days after last drug administration
Number of patients with clinically significant findings in vital signs | up to 5 days after last drug administration
  pulse rate, blood pressure
Number of patients with clinically significant findings in laboratory tests | up to 5 days after last drug administration
Trough concentration of BIBV 308 SE before doses | up to 84 hours